CLINICAL TRIAL: NCT00983372
Title: A One-Directional, Open-Label Drug Interaction Study to Investigate the Effects of Multiple-Dose Diltiazem ER on Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between Colchicine and Diltiazem ER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1015
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Healthy; Adult; Volunteer; Colchicine; Pharmacokinetics; Diltiazem; Cytochrome p450 3A4; P-glycoprotein
Keywords: healthy; adult; volunteer; colchicine; diltiazem; blood levels over time
MeSH Terms: interventions — Colchicine; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): -colchicine baseline pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with steady-state Diltiazem (Experimental): -colchicine pharmacokinetics in presence of steady-state diltiazem
  Interventions: Drug: Diltiazem ER; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone at 7:15 am on Day 1 after an overnight fast of at least 10 hours.
  Other Names: COLCRYS™
  Arms: Colchicine alone
Drug: Diltiazem ER — One 240 mg diltiazem ER capsule administered daily at 7:15 am on Days 15 to 21.
  Other Names: Cardizem® CD (Biovail Pharmaceuticals, Inc.)
  Arms: Colchicine with steady-state Diltiazem
Drug: Colchicine — A single dose of 0.6 mg colchicine administered along with diltiazem ER at 7:15 am on Day 21 after an overnight fast of at least 10 hours.
  Arms: Colchicine with steady-state Diltiazem

SUMMARY:
Colchicine is a substrate for both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp). Extended-release diltiazem (diltiazem ER) is a potent inhibitor of both CYP3A4 and P-gp. This study will evaluate the effect of multiple doses of diltiazem ER on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Colchicine is a substrate for both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp). Extended-release diltiazem (diltiazem ER) is a potent inhibitor of both CYP3A4 and P-gp. This study will evaluate the effect of multiple doses of diltiazem ER on the pharmacokinetic profile of a single 0.6mg dose of colchicine. On Day 1 after a fast of at least 10 hours, twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given a single oral dose of colchicine (1 x 0.6 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for twenty-four hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will then continue on a non-confined basis at 36, 48, 72, and 96 hours post-dose. After a 14-day washout period, beginning on Day 15 and continuing through Day 20 all subjects will return to the clinic for non-confined dosing of diltiazem ER (1 x 240 mg capsule daily). Administered diltiazem ER doses on these days will not necessarily be in a fasted state. On Day 21 after a fast of at least 10 hours, all study participants will receive a co-administered single oral dose of colchicine (1 x 0.6 mg tablet) and diltiazem ER (1 x 240 mg capsule). Blood samples will be drawn from all participants before dosing and for twenty-four hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine in the presence of diltiazem ER at steady state. Blood sampling will then continue on a non-confined basis at 36, 48, 72, and 96 hours post-dose administration. Fasting will continue for 4 hours following the co-administered dose of colchicine and diltiazem ER. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (blood pressure and pulse) will be measured pre-dose and at 1, 2, and 3 hours post-dosing on Day 1, pre-dose and 12 hours post-dosing on Day 15 (subjects will return to the study center for the 12-hour post-dose vital sign measurements), and pre-dose and 1, 2, 3 and 12 hours post-dosing on Day 21 to coincide with peak plasma concentrations of both colchicine and diltiazem. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive.

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine or diltiazem.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, PharmD, Principal Investigator — PRACS - Cetero
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking , male and female volunteers, consisting of members of the community at large, were enrolled in the study.
Pre-assignment Details: 53 subjects were screened, 13 were screen failures, 14 had schedule conflicts, 1 transferred to a different study, and 1 was not needed
Groups:
- Colchicine Alone / With Diltiazem (at Steady-state): [All subjects received each of the study treatments.] Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast of at least 10 hours, followed by a washout period of 14 days. On Days 15 to 20, each subject received one 240 mg diltiazem ER capsule at 7:15 a.m. Then, on Day 21, each subject received both one 0.6 mg colchicine tablet and one 240 mg diltiazem ER capsule at 7:15 a.m. after an overnight fast of at least 10 hours.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Diltiazem (at Steady-state)
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone / With Diltiazem (at Steady-state)
Started | 24
Completed | 23 (subject withdrew consent due to schedule conflict - during washout period or diltiazem alone)
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Diltiazem ER Alone
Arm/Group | Colchicine Alone / With Diltiazem (at Steady-state)
Started | 23
Completed | 20 (two subjects dropped due to missed diltiazem ER dose; one subject dropped due to vomitting)
Not Completed | 3
Not completed — missed diltiazem dose | 2
Not completed — Adverse Event | 1
Period: Colchicine With Diltiazem ER
Arm/Group | Colchicine Alone / With Diltiazem (at Steady-state)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone / With Diltiazem (at Steady-state)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to dosing on Days 1 and 21, and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 hours after dose administration
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast of at least 10 hours, followed by a washout period of 14 days.
- Colchicine With Diltiazem (at Steady-state): On Days 15 to 20, each subject received one 240 mg diltiazem ER capsule at 7:15 a.m. Then, on Day 21, each subject received both one 0.6 mg colchicine tablet and one 240 mg diltiazem ER capsule at 7:15 a.m. after an overnight fast of at least 10 hours.
Arm/Group | Colchicine Alone | Colchicine With Diltiazem (at Steady-state)
Number analyzed (Participants) | 20 | 20
pg/mL | 2,172.32 (868.72) | 2,802.90 (1,245.01)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Diltiazem (at Steady-state)
Number analyzed (Participants) | 20 | 20
pg-hr/mL | 10,035.57 (4,562.57) | 17,729.64 (8,642.59)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Diltiazem (at Steady-state)
Number analyzed (Participants) | 20 | 20
pg-hr/mL | 12,025.69 (5,418.95) | 22,485.97 (10,994.16)

ADVERSE EVENTS:
Groups:
- Diltiazem Alone: On Days 15 to 20, each subject received one 240 mg diltiazem ER capsule at 7:15 a.m.
- Colchicine With Steady-state Diltiazem: On Day 21, each subject received both one 0.6 mg colchicine tablet and one 240 mg diltiazem ER capsule at 7:15 a.m. after an overnight fast of at least 10 hours.
Arm/Group | Colchicine Alone | Diltiazem Alone | Colchicine With Steady-state Diltiazem
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 6 | 9 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Diltiazem Alone | Colchicine With Steady-state Diltiazem
dry eye (Eye disorders) | 1/24 (1) | 0/21 (0) | 0/20 (0)
eye irritation (Eye disorders) | 1/24 (1) | 0/21 (0) | 0/20 (0)
dyspepsia (Gastrointestinal disorders) | 0/24 (0) | 1/21 (1) | 0/20 (0)
nausea (Gastrointestinal disorders) | 1/24 (1) | 1/21 (1) | 1/20 (1)
vomiting (Gastrointestinal disorders) | 0/24 (0) | 1/21 (1) | 0/20 (0)
chest pain (General disorders) | 1/24 (1) | 0/21 (0) | 0/20 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/24 (1) | 0/21 (0) | 0/20 (0)
dizziness (Nervous system disorders) | 0/24 (0) | 1/21 (1) | 0/20 (0)
headache (Nervous system disorders) | 2/24 (2) | 8/21 (11) | 3/20 (3)
lethargy (Nervous system disorders) | 0/24 (0) | 0/21 (0) | 1/20 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/24 (1) | 0/21 (0) | 0/20 (0)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 0/21 (0) | 1/20 (2)
contact dermatitis (Skin and subcutaneous tissue disorders) | 0/24 (0) | 1/21 (1) | 0/20 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days